CLINICAL TRIAL: NCT01371162
Title: A Multi-Center, Randomized, Double-Blind, Multiple Ascending Dose, Placebo-Controlled, Parallel Group 2-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic of the HCV Nucleoside Inhibitor RO5428029 in Healthy Subjects and in CHC Genotype 1 Infected Patients
Brief Title: A Study of RO5428029 in Healthy Volunteers and Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NP25733
Record Dates: First submitted 2011-06-06; First posted 2011-06-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic, Healthy Volunteer
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A1 Healthy Volunteers (Experimental)
  Interventions: Drug: RO5428029
- A2 (Placebo Comparator)
  Interventions: Drug: placebo
- B1 HCV Infection (Experimental)
  Interventions: Drug: RO5428029
- B2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RO5428029 — Multiple ascending doses
  Arms: A1 Healthy Volunteers; B1 HCV Infection
Drug: placebo — multiple doses
  Arms: A2; B2

SUMMARY:
This 2-part, randomized, double-blind, placebo-controlled study will assess the safety, pharmacokinetics and pharmacodynamics of RO5428029 in healthy volunteers and patients with hepatitis C infection. Cohorts will be randomized to receive either RO5428029 in ascending doses or placebo for up to 7 days (patients) or up to 14 days (healthy volunteers).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (Part A) or patients with chronic hepatitis C infection (Part B), 18 to 60 years of age, inclusive
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive, and a minimum weight of 45 kg
* Female subjects/patients must be surgically sterile or post-menopausal
* Male subjects/patients and their partners of childbearing potential must use 2 methods of contraception
* For HCV patients:
* Hepatitis C genotype 1 of > 6 months duration at screening
* HCV RNA quantifiable (Roche COBAS TaqMan HCV Test) at screening
* HCV treatment-naïve (no prior antiviral therapy for chronic hepatitis C with interferon-based therapy)
* Liver biopsy or non-invasive procedure within the past 2 years showing absence of cirrhosis

Exclusion Criteria:

* Pregnant or lactating women, and male partners of women who are pregnant or lactating
* Positive test for drugs of abuse
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams or 1 unit of alcohol
* History or symptoms of any significant disease or disorder
* History of active malignancy within the last 5 years, except for localized or in situ carcinoma (e.g. basal or squamous cell carcinoma of the skin)
* Positive for hepatitis B or HIV infection, and/ or for HCV for healthy volunteers (Part A)
* For HCV patients:
* Decompensated liver disease or impaired liver function as defined by any history of ascites, hepatic encephalopathy, hepatocellular carcinoma or bleeding esophageal varices, or prothrombin international normalized ratio (PTINR) >/= 2.0 at screening
* Evidence of cirrhosis and/or incomplete transition to cirrhosis
* Presence or history of non-hepatitis C liver disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Part B: Viral load response: HCV RNA (assessed by Roche COBAS Taqman HCV Test) | up to 17 days
Parts A + B: Safety: Incidence of adverse events | up to 24 days
Parts A + B: Pharmacokinetics: Area under the concentration - time curve (AUC) | up to 24 days

SECONDARY OUTCOMES:
Part B: Viral resistance (viral breakthrough/non-response/partial response) HCV RNA assessed by Roche COBAS Paqman HCV Test | up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- France (2):
  - Montpellier
  - Strasbourg
- Leiden, Netherlands
- Poland (3):
  - Chorzów
  - Warsaw
  - Wroclaw